CLINICAL TRIAL: NCT01774669
Title: Effectiveness of the YouGrabber System Using Virtual Reality in Stroke Rehabilitation: a Single Blinded, Randomised Controlled Multi-centre Trial
Brief Title: Effectiveness Study on a Virtual Reality Based Training System for Stroke Patients
Acronym: YouGrabber
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reha Rheinfelden (Other)
Collaborators: YouRehab Inc. (Industry); Swiss Commission for Technology and Innovation (Other)
Responsible Party: Principal Investigator, PD Dr. Daniel Kiper, Principal Investigator, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/065; 220/12 (Other: Ethics committee Bern)
Record Dates: First submitted 2013-01-15; First posted 2013-01-24 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2015-11

CONDITIONS: Cerebrovascular Accident; Hemorrhagic Stroke; Stroke
Keywords: ischemic stroke; hemorrhagic stroke; upper limb; virtual reality; physiotherapy; occupational therapy
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke; Ischemic Stroke | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- YouGrabber training device from YouRehab Ltd. (Experimental): Patients in the experimental group (EG) will receive 16 training sessions lasting for 45 minutes each.
  Interventions: Device: YouGrabber training device from YouRehab Ltd.
- Conventional therapy (Active Comparator): Patients in the control group (CG) will receive 16 therapy sessions (physiotherapy or occupational therapy) lasting for 45 minutes each.
  Interventions: Other: Therapy (PT, OT)

INTERVENTIONS:
Device: YouGrabber training device from YouRehab Ltd. — Patients in the experimental group (EG) will receive 16 training sessions lasting for 45 minutes each. The treatment focus is the upper extremity, in particular finder and hand function, movement coordination, and speed.
  Arms: YouGrabber training device from YouRehab Ltd.
Other: Therapy (PT, OT) — Patients in the control group (CG) will receive 16 therapy sessions physiotherapy or occupational therapy) lasting for 45 minutes each. The therapy focuses on upper limb movements, in particular finger and hand movements. Furthermore, movement coordination and speed shall be trained.
  Arms: Conventional therapy

SUMMARY:
The patient study is a phase III trial designed as a single-blinded, randomised, controlled multi-centre trial with repeated measurement events (ME). Patients will be evaluated by a blinded assessor on five occasions: twice within two weeks at baseline before intervention start (BL, T0), once after eight treatment sessions (T1), once after the intervention (T2), and once after a two month follow-up period (FU). Figure 1 illustrates the study overview.

The study focuses on the evaluation of the YouGrabber efficacy compared to conventional therapy in an outpatient setting.

Research question: Do patients after stroke in the YouGrabber training group show higher postintervention performance in the Box and Block Test (BBT) compared to patients in the conventional therapy group? Hypothesis: H0: The investigators hypothesise that there will be no group differences after 16 training sessions or after the two month follow-up period.

H1: The investigators hypothesise that there will be a group difference after the 16 training sessions and after the two month follow-up period.

Aim: The aim of the project is to design and implement a single-blinded, randomised controlled multi-centre trial comparing YouGrabber training and conventional therapy in patients after stroke.

Patients will be randomly allocated to either the experimental group (EG) or the control group (CG) after the second ME (T0). Group allocation will be based on a computer-generated randomisation list (one for each centre, (MATLAB, 2007b, Mathworks Inc., USA) created by a researcher not involved into the study. Randomisation lists and corresponding token will be stored in the clinics' pharmacy. Patients will draw a token before the first therapy session. The token will be marked and stored until study finalisation in the pharmacy.

Group allocation will remain concealed for the independent assessor until study finalisation. Patients and treating therapists will be reminded not to talk about patient's group allocation with other therapists or participants.

Patients in both study groups (EG, CG) will receive the same amount of 16 sessions lasting for 45 minutes each. During each therapy appointment patients can decide to stop the training at any time.

Patients allocated to EG will have the opportunity to participate in two semi-structured interviews to evaluate their expectations and experiences with the virtual reality therapy with YouGrabber.

Treating therapists will have the opportunity to participate in one focus group meeting to evaluate their experiences with the virtual reality training, its advantages and disadvantages. Interview and focus group participation will be voluntary.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 months after first-ever stroke (ischemic, haemorrhagic)
* Able to sit in a normal chair without armrests and without support of the back rest
* Persistent motor deficit of the arm and hand confirmed by the Chedoke-McMaster Stroke Assessment (CMSA) subscale arm level 7>x=/>3 and subscale hand level 7>x=/>2.

Exclusion Criteria:

* Previous or current other functional deficits of arm and hand motor function not due to stroke.
* Severe cognitive deficits MMSE ≤ 20.
* Severe spatial-visual disorders, e.g. severe visual neglect confirmed by a Line-Bisection-Test.
* History of epileptic seizures triggered by visual stimuli (e.g. television, video games) within the last six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Box and Block Test (BBT) | 15 months
  Patients will be evaluated by a blinded assessor on five occasions: twice within two weeks at baseline before intervention start (BL, T0), once after eight treatment sessions (T1), once after the intervention (T2), and once after a two month follow-up period (FU).

SECONDARY OUTCOMES:
Chedoke-McMaster Stroke Assessment (CMSA) | 15 months
  Patients will be evaluated by a blinded assessor on five occasions: twice within two weeks at baseline before intervention start (BL, T0), once after eight treatment sessions (T1), once after the intervention (T2), and once after a two month follow-up period (FU).
Chedoke Arm and Hand Activity Inventory (CAHAI) | 15 months
  Patients will be evaluated by a blinded assessor on five occasions: twice within two weeks at baseline before intervention start (BL, T0), once after eight treatment sessions (T1), once after the intervention (T2), and once after a two month follow-up period (FU).
Stroke Impact Scale (SIS) | 15 months
  Patients will be evaluated by a blinded assessor on five occasions: twice within two weeks at baseline before intervention start (BL, T0), once after eight treatment sessions (T1), once after the intervention (T2), and once after a two month follow-up period (FU).

OTHER OUTCOMES:
active range of motion (ROM) | 15 months
  Patients will be evaluated by a blinded assessor on five occasions: twice within two weeks at baseline before intervention start (BL, T0), once after eight treatment sessions (T1), once after the intervention (T2), and once after a two month follow-up period (FU).
Extended Barthel Index (EBI) | 15 months
Mini Mental State Examination (MMSE) | 15 months
Edinburgh Handedness Inventory (EHI) | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kiper, PD PhD, Principal Investigator — University and ETH Zurich, Institute for Neuroinformatics
Locations (2):
- Switzerland (2):
  - Reha Rheinfelden, Rheinfelden, Canton of Aargau
  - Inselspital Bern, Bern, Canton of Bern

REFERENCES:
- [Derived] Schuster-Amft C, Eng K, Suica Z, Thaler I, Signer S, Lehmann I, Schmid L, McCaskey MA, Hawkins M, Verra ML, Kiper D. Effect of a four-week virtual reality-based training versus conventional therapy on upper limb motor function after stroke: A multicenter parallel group randomized trial. PLoS One. 2018 Oct 24;13(10):e0204455. doi: 10.1371/journal.pone.0204455. eCollection 2018. PMID 30356229
- [Derived] Schuster-Amft C, Eng K, Lehmann I, Schmid L, Kobashi N, Thaler I, Verra ML, Henneke A, Signer S, McCaskey M, Kiper D. Using mixed methods to evaluate efficacy and user expectations of a virtual reality-based training system for upper-limb recovery in patients after stroke: a study protocol for a randomised controlled trial. Trials. 2014 Sep 6;15:350. doi: 10.1186/1745-6215-15-350. PMID 25194928
- See also: Home page of participating cite. — http://www.reha-rheinfelden.ch/